CLINICAL TRIAL: NCT00654745
Title: A Prospective, Open-label, Ambulatory Blood Pressure Monitoring (ABPM) Dose Titration Study to Evaluate the Safety and Efficacy of an Olmesartan Medoxomil and Amlodipine Based Treatment Regimen in Hypertensive, Type 2 Diabetic Subjects
Brief Title: 18 Week Study Evaluating Safety and Efficacy of Olmesartan, Amlodipine, and Hydrochlorothiazide, in Type 2 Diabetics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Director, Medical Research, Hypertension, Daiichi Sankyo Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-8663-403
Record Dates: First submitted 2008-04-04; First posted 2008-04-09 (Estimated); Results first posted 2010-07-02 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2010-07

CONDITIONS: Type 2 Diabetes; Hypertension
Keywords: blood pressure reduction
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension | interventions — Amlodipine; Amlodipine Besylate, Olmesartan Medoxomil Drug Combination; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- aml + olm + hctz (Experimental): amlodipine; and olmesartan medoxomil, if required; and hydrochlorothiazide, if required.
  Interventions: Drug: Amlodipine; Drug: amlodipine / olmesartan medoxomil combination; Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Amlodipine — Amlodipine 5 mg tablets , Daily for 3 weeks;
  Other Names: Norvasc
Drug: amlodipine / olmesartan medoxomil combination — amlodipine / olmesartan medoxomil combination tablets 5 mg/20 mg or 5 mg/40 mg or 10 mg/40 mg
  Other Names: Azor
Drug: Hydrochlorothiazide — hydrochlorothiazide tablets, 12.5 mg or 25 mg.

SUMMARY:
To determine if olmesartan plus amlodipine combination therapy alone and with hydrochlorothiazide will be safe and effective to reduce high blood pressure in hypertensive, type 2 diabetic subjects.

DETAILED DESCRIPTION:
This is a single group study in which participants were titrated to the next of 6 regimens if blood pressure (BP) goals were not met.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 to 80 years.
* Diagnosis of type 2 diabetes mellitus and on a stable regimen of any oral antidiabetic agent(s) for at least 3 months, with or without adjunctive use of Byetta (exenatide);

Note: Subjects diagnosed with type 2 diabetes mellitus who were not on oral antidiabetic agents may have been enrolled if they had a documented history of type 2 diabetes by American Diabetes Association criteria, including the specific plasma glucose results listed below:

* Fasting plasma glucose >=126 mg/dL (7.0 mmol/L); or
* Symptoms of hyperglycemia and a casual (any time of day without regard to time since last meal) plasma glucose >=200 mg/dL (11.1 mmol/L). The classic symptoms of hyperglycemia were considered to include polyuria, polydipsia, and unexplained weight loss; or
* Two-hour plasma glucose >=200 mg/dL (11.1 mmol/L) during an oral glucose tolerance test;
* Newly diagnosed hypertension or uncontrolled hypertension (defined as SBP >130 mmHg and/or DBP >80 mmHg) on current antihypertensive monotherapy or combination therapy.
* Subjects must fulfill mean seated office blood pressure parameters at two consecutive, qualifying visits during the placebo run-in phase, and, subsequently, daytime ambulatory blood pressure monitoring (ABPM) criteria.
* Females should not be pregnant or lactating and, if applicable, using adequate contraception.

Exclusion Criteria:

* Subjects with uncontrolled hypertension taking multiple antihypertensive therapies (at the discretion of the investigator).
* Type 2 diabetes mellitus with a glycosylated hemoglobin A1c (HbA1c) >=9.0% at screening;
* Subjects with type 1 or type 2 diabetes mellitus requiring insulin.
* Subjects with any serious disorder which may limit the ability to evaluate the safety and efficacy of study medication, or subjects with secondary hypertension.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2008-05; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Los Angeles, California
  - Sylmar, California
  - Tustin, California
  - Aventura, Florida
  - DeLand, Florida
  - Hialeah, Florida
  - Pembroke Pines, Florida
  - Avon, Indiana
  - Indianapolis, Indiana
  - Las Vegas, Nevada
  - New Windsor, New York
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Charleston, South Carolina
  - Greer, South Carolina
  - Taylors, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - Burke, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at 32 sites in the USA from May 12, 2008 to Jan 2, 2009 and 207 enrolled into the active treatment period. The study population consisted of subjects with controlled type 2 diabetes, not requiring insulin therapy, whose hypertension was newly diagnosed or uncontrolled on antihypertensive monotherapy or combination therapy.
Pre-assignment Details: Subjects began washout of anti-hypertensive medications during screening then entered placebo run-in lasting 2-3 weeks. Subjects must meet seated blood pressure (BP) criteria at 2 consecutive qualifying visits during the run-in period and satisfy mean daytime ambulatory BP criteria at baseline, one day prior to the first dose of active study drug.
Groups:
- Amlodipine, Olmesartan Medoxomil, Hydrochlorothiazide: Participants receiving amlodipine + olmesartan medoxomil, if required, + hydrochlorothiazide, if required
Period: Overall Study
Arm/Group | Amlodipine, Olmesartan Medoxomil, Hydrochlorothiazide
Started | 207 (This is single group study in which subjects were titrated to the next of 7 arms if BP goal not met.)
Completed | 164
Not Completed | 43
Not completed — Adverse Event | 12
Not completed — Lost to Follow-up | 7
Not completed — Protocol Violation | 11
Not completed — Withdrawal by Subject | 10
Not completed — poor ABPM, noncompliance, lab MAs | 3

BASELINE CHARACTERISTICS:
Groups:
- Aml + Olm + Hctz: amlodipine (aml) + olmesartan medoxomil (olm)+ hhdrochlorothiazide (hctz) is total number enrolled. Each group is the number of participants that were titrated to that dosing regimen as per the protocol. The total number of participants of the individual groups does not (and should not) equal the total number enrolled.
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 207
Age Continuous [Mean (Standard Deviation); unit: years] | 59.1 (9.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122
  Male | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54
  Not Hispanic or Latino | 153
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 35
  White | 162
  More than one race | 0
  Unknown or Not Reported | 0
Stage of hypertension [Number; unit: participants] — Stage 1 or Stage 2 Hypertension. Stage 1 = Blood pressure > 140/90 mm Hg. Stage 2 = systolic >160 mm Hg or diastolic > 100 mm Hg
  participants
    Stage 1 | 115
    Stage 2 | 92
Body mass index [Mean (Standard Deviation); unit: mg/m2] | 32.80 (5.947)
Mean 24-hour ambulatory diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 81.6 (9.76)
Mean 24-hour ambulatory systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 144.4 (11.74)
Pulse rate [Mean (Standard Deviation); unit: beats per minute] | 73.75 (11.909)
Seated Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 89.1 (10.13)
Seated Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 158.8 (13.14)
Years with diabetes [Mean (Standard Deviation); unit: years] | 6.44 (5.978)

OUTCOME MEASURES:

1. Primary Outcome: Change From Week 0 (Baseline) in Mean 24-hour Ambulatory Blood Pressure Monitoring (ABPM) Systolic Blood Pressure (SBP) After 12 Weeks of Active Treatment
Description: Change from week 0 (baseline) in mean 24-hour Ambulatory Blood Pressure Monitoring (ABPM) Systolic Blood Pressure (SBP) after 12 weeks of active treatment. change = week 12 - week 0.
Time Frame: week 0 - week 12
Population: ABPM subjects analysis population included 165 subjects who received at least one dose of active study medication and provided valid ambulatory blood pressure monitoring measurements at baseline and week 12.
Measure: Mean (Standard Error); unit: mm Hg
Groups:
- Aml + Olm + Hctz: amlodipine + olmesartan medoxomil, if required, + hydrochlorothiazide, if required
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 165
mm Hg | -19.9 (0.76)
Statistical Analysis 1: Comparison: Aml + Olm + Hctz; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Net) = -19.9, 95% CI 2-sided [-21.5 to -18.4]

2. Secondary Outcome: Change From Week 0 (Baseline) in Mean ABPM Diastolic Blood Pressure (DBP) After 12 Weeks of Active Treatment
Description: 24-hour mean DBP, Daytime mean DBP, Nighttime mean DBP, Last 6 hour mean DBP, Last 4 hour mean DBP, Last 2 hour mean DBP
Time Frame: week 0 - week 12 (24-hour, Daytime, Nighttime, Last 6 hour, Last 4 hour, Last 2 hour)
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 165
mm Hg
  24-hour mean DBP change from baseline | -11.2 (0.50)
  daytime mean DBP change from baseline | -11.7 (0.60)
  nighttime mean DBP change from baseline | -10.4 (0.68)
  last 6 hour mean DBP change from baseline | -10.9 (0.64)
  last 4 hour mean DBP change from baseline | -11.1 (0.68)
  last 2 hour mean DBP change from baseline | -11.5 (0.76)
Statistical Analysis 1: Comparison: Aml + Olm + Hctz; Primary null hypothesis is change from baseline to week12 in ABPM is 0. Change from baseline to week12 is primary efficacy variable and used all ABPM subjects. Null hypothesis used 1-sample t-test on change. Sample size of 200 expected to provide 99% power at significance level of 0.05%; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — 24-hour mean DBP change from baseline to week 12; standard 1-sample confidence interval construction using t-distribution with 164 degrees of freedom; Mean Difference (Net) = -11.2, 95% CI 2-sided [-12.2 to -10.3]
Statistical Analysis 2: Comparison: Aml + Olm + Hctz; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — daytime mean DBP change from baseline to week 12; standard 1-sample confidence interval construction using t-distribution with 164 degrees of freedom; Mean Difference (Net) = -11.7, 95% CI 2-sided [-12.9 to -10.5]
Statistical Analysis 3: Comparison: Aml + Olm + Hctz; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — nighttime mean DBP change from baseline to week 12; standard 1-sample confidence interval construction using t-distribution with 164 degrees of freedom; Mean Difference (Net) = -10.4, 95% CI 2-sided [-11.7 to -9.0]
Statistical Analysis 4: Comparison: Aml + Olm + Hctz; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — last 6 hours mean DBP change from baseline to week 12; standard 1-sample confidence interval construction using t-distribution with 164 degrees of freedom; Mean Difference (Net) = -10.9, 95% CI 2-sided [-12.2 to -9.7]
Statistical Analysis 5: Comparison: Aml + Olm + Hctz; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — last 4 hours mean DBP change from baseline to week 12; standard 1-sample confidence interval construction using t-distribution with 164 degrees of freedom; Mean Difference (Net) = -11.1, 95% CI 2-sided [-12.4 to -9.8]
Statistical Analysis 6: Comparison: Aml + Olm + Hctz; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — last 2 hours mean DBP change from baseline to week 12; standard 1-sample confidence interval construction using t-distribution with 164 degrees of freedom; Mean Difference (Net) = -11.5, 95% CI 2-sided [-13.1 to -10.0]

3. Secondary Outcome: Change From Week 0 (Baseline) in Mean ABPM SBP After 12 Weeks of Active Treatment
Description: Daytime mean SBP, Nighttime mean SBP, Last 6 hour mean SBP, Last 4 hour mean SBP, Last 2 hour mean SBP
Time Frame: week 0 - week 12 (24-hour, Daytime, Nighttime, Last 6 hour, Last 4 hour, Last 2 hour)
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 165
mm Hg
  daytime mean SBP change from baseline | -20.8 (0.92)
  nighttime mean SBP change from baseline | -18.5 (0.95)
  last 6 hours mean SBP change from baseline | -18.9 (0.93)
  last 4 hours mean SBP change from baseline | -19.1 (1.02)
  last 2 hours mean SBP change from baseline | -19.5 (1.10)
Statistical Analysis 1: Comparison: Aml + Olm + Hctz; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — daytime mean SBP change from baseline to week 12; standard 1-sample confidence interval construction using t-distribution with 164 degrees of freedom; Mean Difference (Net) = -20.8, 95% CI 2-sided [-22.6 to -18.9]
Statistical Analysis 2: Comparison: Aml + Olm + Hctz; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — nighttime mean SBP change from baseline to week 12; standard 1-sample confidence interval construction using t-distribution with 164 degrees of freedom; Mean Difference (Net) = -18.5, 95% CI 2-sided [-20.4 to -16.6]
Statistical Analysis 3: Comparison: Aml + Olm + Hctz; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — last 6 hours mean SBP change from baseline to week 12; standard 1-sample confidence interval construction using t-distribution with 164 degrees of freedom; Mean Difference (Net) = -18.9, 95% CI 2-sided [-20.7 to -17.0]
Statistical Analysis 4: Comparison: Aml + Olm + Hctz; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — last 4 hours mean SBP change from baseline to week 12; standard 1-sample confidence interval construction using t-distribution with 164 degrees of freedom; Mean Difference (Net) = -19.1, 95% CI 2-sided [-21.1 to -17.1]
Statistical Analysis 5: Comparison: Aml + Olm + Hctz; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — last 2 hours mean SBP change from baseline to week 12; standard 1-sample confidence interval construction using t-distribution with 164 degrees of freedom; Mean Difference (Net) = -19.5, 95% CI 2-sided [-21.7 to -17.4]

4. Secondary Outcome: Change in Mean Seated Systolic Blood Pressure (SeSBP) From Week 0 (Baseline) After 3, 6, 9, 12, 15, and 18 Weeks
Description: change in mean SeSBP from week 0 (baseline) to Weeks 3, 6, 9, 12, 15, and 18.
Time Frame: week 0 - weeks 3, 6, 9, 12, 15, 18
Population: Number of participants changed by week. Week 3 = 201, Week 6 = 192, week 9 = 184, week 12 = 177, week 15 = 172, week 18 = 164.
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 201
mm Hg
  week 3 mean SBP change from baseline | -10.3 (0.87)
  week 6 mean SBP change from baseline | -17.9 (0.92)
  week 9 mean SBP change from baseline | -20.0 (1.10)
  week 12 mean SBP change from baseline | -23.7 (1.02)
  week 15 mean SBP change from baseline | -28.5 (1.16)
  week 18 mean SBP change from baseline | -31.1 (1.13)
Statistical Analysis 1: Comparison: Aml + Olm + Hctz; Primary null hypothesis is change from baseline is 0. Null hypothesis used 1-sample t-test on change. Sample size of 200 expected to provide 99% power at significance level of 0.05%; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Change in mean seated systolic blood pressure from baseline to week 3; standard 1-sample confidence interval construction using t-distribution with n-1 degrees of freedom; Mean Difference (Net) = -10.3, 95% CI 2-sided [-12.0 to -8.6]
Statistical Analysis 2: Comparison: Aml + Olm + Hctz; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Change in mean seated systolic blood pressure from baseline to week 6; standard 1-sample confidence interval construction using t-distribution with n-1 degrees of freedom; Mean Difference (Net) = -17.9, 95% CI 2-sided [-19.8 to -16.1]
Statistical Analysis 3: Comparison: Aml + Olm + Hctz; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Change in mean seated systolic blood pressure from baseline to week 9; standard 1-sample confidence interval construction using t-distribution with n-1 degrees of freedom; Mean Difference (Net) = -20.0, 95% CI 2-sided [-22.2 to -17.8]
Statistical Analysis 4: Comparison: Aml + Olm + Hctz; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Change in mean seated systolic blood pressure from baseline to week 12; standard 1-sample confidence interval construction using t-distribution with n-1 degrees of freedom; Mean Difference (Net) = -23.7, 95% CI 2-sided [-25.7 to -21.7]
Statistical Analysis 5: Comparison: Aml + Olm + Hctz; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Change in mean seated systolic blood pressure from baseline to week 15; standard 1-sample confidence interval construction using t-distribution with n-1 degrees of freedom; Mean Difference (Net) = -28.5, 95% CI 2-sided [-30.8 to -26.2]
Statistical Analysis 6: Comparison: Aml + Olm + Hctz; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Change in mean seated systolic blood pressure from baseline to week 18; standard 1-sample confidence interval construction using t-distribution with n-1 degrees of freedom; Mean Difference (Net) = -31.1, 95% CI 2-sided [-33.3 to -28.8]

5. Secondary Outcome: Change in Mean Seated Diastolic Blood Pressure (SeDBP) From Week 0 (Baseline) After 3, 6, 9, 12, 15, and 18 Weeks
Description: change in mean SeDBP from week 0 (baseline) to Weeks 3, 6, 9, 12, 15, and 18.
Time Frame: week 0 - weeks 3, 6, 9, 12, 15, 18
Population: as for outcome 4
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 201
mm Hg
  week 3 mean seDBP change from baseline | -4.1 (0.50)
  week 6 mean seDBP change from baseline | -8.2 (0.60)
  week 9 mean seDBP change from baseline | -9.7 (0.64)
  week 12 mean seDBP change from baseline | -11.2 (0.64)
  week 15 mean seDBP change from baseline | -14.4 (0.66)
  week 18 mean seDBP change from baseline | -15.1 (0.72)
Statistical Analysis 1: Comparison: Aml + Olm + Hctz; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Change in mean seated diastolic blood pressure from baseline to week 3; standard 1-sample confidence interval construction using t-distribution with n-1 degrees of freedom; Mean Difference (Net) = -4.1, 95% CI 2-sided [-5.1 to -3.1]
Statistical Analysis 2: Comparison: Aml + Olm + Hctz; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Change in mean seated diastolic blood pressure from baseline to week 6; standard 1-sample confidence interval construction using t-distribution with n-1 degrees of freedom; Mean Difference (Net) = -8.2, 95% CI 2-sided [-9.4 to -7.1]
Statistical Analysis 3: Comparison: Aml + Olm + Hctz; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Change in mean seated diastolic blood pressure from baseline to week 9; standard 1-sample confidence interval construction using t-distribution with n-1 degrees of freedom; Mean Difference (Net) = -9.7, 95% CI 2-sided [-10.9 to -8.4]
Statistical Analysis 4: Comparison: Aml + Olm + Hctz; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Change in mean seated diastolic blood pressure from baseline to week 12; standard 1-sample confidence interval construction using t-distribution with n-1 degrees of freedom; Mean Difference (Net) = -11.2, 95% CI 2-sided [-12.5 to -9.9]
Statistical Analysis 5: Comparison: Aml + Olm + Hctz; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Change in mean seated diastolic blood pressure from baseline to week 15; standard 1-sample confidence interval construction using t-distribution with n-1 degrees of freedom; Mean Difference (Net) = -14.4, 95% CI 2-sided [-15.7 to -13.1]
Statistical Analysis 6: Comparison: Aml + Olm + Hctz; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Change in mean seated diastolic blood pressure from baseline to week 18; standard 1-sample confidence interval construction using t-distribution with n-1 degrees of freedom; Mean Difference (Net) = -15.1, 95% CI 2-sided [-16.5 to -13.6]

6. Secondary Outcome: Number of Participants Achieving Mean 24-hour Ambulatory Blood Pressure Thresholds at Week 12
Description: number of participants achieving mean 24-hour ambulatory blood pressure thresholds BP<135/85, BP<130/80, BP<125/75, BP<120/80, SBP<135, SBP<130, SBP<125, SBP<120, DBP<85, DBP<80, DBP<75 at week 12
Time Frame: week 0 - week 12
Measure: Number; unit: participants
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 165
participants
  mean 24-hour BP <135/85 | 140
  mean 24-hour BP <130/80 | 116
  mean 24-hour BP <125/75 | 76
  mean 24-hour BP <120/80 | 59
  mean 24-hour SBP <135 | 140
  mean 24-hour SBP <130 | 120
  mean 24-hour SBP <125 | 92
  mean 24-hour SBP <120 | 59
  mean 24-hour DBP <85 | 158
  mean 24-hour DBP <80 | 146
  mean 24-hour DBP <75 | 121

7. Secondary Outcome: Number of Participants Achieving Mean Daytime Ambulatory Blood Pressure Thresholds at Week 12
Description: number of participants achieving mean daytime ambulatory blood pressure thresholds BP<135/85, BP<130/80, BP<125/75, BP<120/80, SBP<135, SBP<130, SBP<125, SBP<120, DBP<85, DBP<80, DBP<75 at week 12
Time Frame: week 0 - week 12
Measure: Number; unit: participants
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 165
participants
  mean daytime BP < 135/85 | 116
  mean daytime BP < 130/80 | 83
  mean daytime BP < 125/75 | 48
  mean daytime BP < 120/80 | 42
  mean daytime SBP < 135 | 118
  mean daytime SBP < 130 | 94
  mean daytime SBP < 125 | 67
  mean daytime SBP < 120 | 42
  mean daytime DBP < 85 | 151
  mean daytime DBP < 80 | 124
  mean daytime DBP < 75 | 91

8. Secondary Outcome: Number of Participants Achieving Mean Nighttime Ambulatory Blood Pressure Thresholds at Week 12
Description: number of participants achieving mean nighttime ambulatory blood pressure thresholds BP<135/85, BP<130/80, BP<125/75, BP<120/80, BP<120/70, SBP<135, SBP<130, SBP<125, SBP<120, DBP<85, DBP<80, DBP<75, DBP<70 at week 12
Time Frame: week 0 - week 12
Measure: Number; unit: participants
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 165
participants
  mean nighttime BP < 135/85 | 152
  mean nighttime BP < 130/80 | 137
  mean nighttime BP < 125/75 | 119
  mean nighttime BP < 120/80 | 112
  mean nighttime BP < 120/70 | 101
  mean nighttime SBP < 135 | 154
  mean nighttime SBP < 130 | 139
  mean nighttime SBP < 125 | 123
  mean nighttime SBP < 120 | 112
  mean nighttime DBP < 85 | 160
  mean nighttime DBP < 80 | 158
  mean nighttime DBP < 75 | 147
  mean nighttime DBP < 70 | 124

9. Secondary Outcome: Number of Participants Achieving Mean Last 6 Hour Ambulatory Blood Pressure Thresholds at Week 12
Description: number participants achieving mean last 6 hour ambulatory blood pressure thresholds BP<135/85, BP<130/80, BP<125/75, BP<120/80, SBP<135, SBP<130, SBP<125, SBP<120, DBP<85, DBP<80, DBP<75 at week 12
Time Frame: week 0 - week 12
Measure: Number; unit: participants
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 165
participants
  mean last 6 hour BP < 135/85 | 135
  mean last 6 hour BP < 130/80 | 124
  mean last 6 hour BP < 125/75 | 101
  mean last 6 hour BP < 120/80 | 85
  mean last 6 hour SBP < 135 | 143
  mean last 6 hour SBP < 130 | 127
  mean last 6 hour SBP < 125 | 108
  mean last 6 hour SBP < 120 | 85
  mean last 6 hour DBP < 85 | 157
  mean last 6 hour DBP < 80 | 146
  mean last 6 hour DBP < 75 | 130

10. Secondary Outcome: Number of Participants Achieving Mean Last 4 Hour Ambulatory Blood Pressure Thresholds at Week 12
Description: number of participants achieving mean last 4 hour ambulatory blood pressure thresholds BP<135/85, BP<130/80, BP<125/75, BP<120/80, SBP<135, SBP<130, SBP<125, SBP<120, DBP<85, DBP<80, DBP<75 at week 12
Time Frame: week 0 - week 12
Measure: Number; unit: participants
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 165
participants
  mean last 4 hour BP < 135/85 | 129
  mean last 4 hour BP < 130/80 | 107
  mean last 4 hour BP < 125/75 | 92
  mean last 4 hour BP < 120/80 | 72
  mean last 4 hour SBP < 135 | 131
  mean last 4 hour SBP < 130 | 114
  mean last 4 hour SBP < 125 | 102
  mean last 4 hour SBP < 120 | 72
  mean last 4 hour DBP < 85 | 150
  mean last 4 hour DBP < 80 | 137
  mean last 4 hour DBP < 75 | 120

11. Secondary Outcome: Number of Participants Achieving Mean Last 2 Hour Ambulatory Blood Pressure Thresholds at Week 12
Description: number of participants achieving mean last 2 hour ambulatory blood pressure thresholds BP<135/85, BP<130/80, BP<125/75, BP<120/80, SBP<135, SBP<130, SBP<125, SBP<120, DBP<85, DBP<80, DBP<75 at week 12
Time Frame: week 0 - week 12
Measure: Number; unit: participants
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 165
participants
  mean last 2 hour BP < 135/85 | 110
  mean last 2 hour BP < 130/80 | 85
  mean last 2 hour BP < 125/75 | 63
  mean last 2 hour BP < 120/80 | 49
  mean last 2 hour SBP < 135 | 115
  mean last 2 hour SBP < 130 | 92
  mean last 2 hour SBP < 125 | 76
  mean last 2 hour SBP < 120 | 51
  mean last 2 hour DBP < 85 | 145
  mean last 2 hour DBP < 80 | 125
  mean last 2 hour DBP < 75 | 94

12. Secondary Outcome: Number of Participants Achieving Seated Systolic and Diastolic Blood Pressure Thresholds at Week 3
Description: number of participants achieving seated systolic and diastolic blood pressure thresholds BP<135/85, BP<130/80, BP<125/75, BP<120/80, SBP<135, SBP<130, SBP<125, SBP<120, DBP<85, DBP<80, DBP<75 at week 3
Time Frame: week 0 - week 3
Measure: Number; unit: participants
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 201
participants
  mean BP < 135/85 | 31
  mean BP < 130/80 | 10
  mean BP < 125/75 | 4
  mean BP < 120/80 | 2
  mean SBP < 135 | 41
  mean SBP < 130 | 17
  mean SBP < 125 | 9
  mean SBP < 120 | 2
  mean DBP < 85 | 99
  mean DBP < 80 | 58
  mean DBP < 75 | 29

13. Secondary Outcome: Number of Participants Achieving Seated Systolic and Diastolic Blood Pressure Thresholds at Week 6
Description: number of participants achieving seated systolic and diastolic blood pressure thresholds BP<135/85, BP<130/80, BP<125/75, BP<120/80, SBP<135, SBP<130, SBP<125, SBP<120, DBP<85, DBP<80, DBP<75 at week 6
Time Frame: week 0 - week 6
Measure: Number; unit: participants
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 192
participants
  mean BP < 135/85 | 61
  mean BP < 130/80 | 36
  mean BP < 125/75 | 18
  mean BP < 120/80 | 13
  mean SBP < 135 | 73
  mean SBP < 130 | 48
  mean SBP < 125 | 31
  mean SBP < 120 | 14
  mean DBP < 85 | 127
  mean DBP < 80 | 91
  mean DBP < 75 | 48

14. Secondary Outcome: Number of Participants Achieving Seated Systolic and Diastolic Blood Pressure Thresholds at Week 9
Description: number of participants achieving seated systolic and diastolic blood pressure thresholds BP<135/85, BP<130/80, BP<125/75, BP<120/80, SBP<135, SBP<130, SBP<125, SBP<120, DBP<85, DBP<80, DBP<75 at week 9
Time Frame: week 0 - week 9
Measure: Number; unit: participants
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 184
participants
  mean BP < 135/85 | 76
  mean BP < 130/80 | 47
  mean BP < 125/75 | 25
  mean BP < 120/80 | 19
  mean SBP < 135 | 82
  mean SBP < 130 | 61
  mean SBP < 125 | 41
  mean SBP < 120 | 20
  mean DBP < 85 | 132
  mean DBP < 80 | 95
  mean DBP < 75 | 64

15. Secondary Outcome: Number of Participants Achieving Seated Systolic and Diastolic Blood Pressure Thresholds at Week 12
Description: number of participants achieving seated systolic and diastolic blood pressure thresholds BP<135/85, BP<130/80, BP<125/75, BP<120/80, SBP<135, SBP<130, SBP<125, SBP<120, DBP<85, DBP<80, DBP<75 at week 12
Time Frame: week 0 - week 12
Measure: Number; unit: participants
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 177
participants
  mean BP < 135/85 | 86
  mean BP < 130/80 | 61
  mean BP < 125/75 | 33
  mean BP < 120/80 | 28
  mean SBP < 135 | 93
  mean SBP < 130 | 70
  mean SBP < 125 | 46
  mean SBP < 120 | 28
  mean DBP < 85 | 134
  mean DBP < 80 | 105
  mean DBP < 75 | 74

16. Secondary Outcome: Number of Participants Achieving Seated Systolic and Diastolic Blood Pressure Thresholds at Week 15
Description: number of participants achieving seated systolic and diastolic blood pressure thresholds BP<135/85, BP<130/80, BP<125/75, BP<120/80, SBP<135, SBP<130, SBP<125, SBP<120, DBP<85, DBP<80, DBP<75 at week 15
Time Frame: week 0 - week 15
Measure: Number; unit: participants
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 172
participants
  mean BP < 135/85 | 114
  mean BP < 130/80 | 83
  mean BP < 125/75 | 51
  mean BP < 120/80 | 45
  mean SBP < 135 | 116
  mean SBP < 130 | 95
  mean SBP < 125 | 69
  mean SBP < 120 | 48
  mean DBP < 85 | 153
  mean DBP < 80 | 122
  mean DBP < 75 | 96

17. Secondary Outcome: Number of Participants Achieving Seated Systolic and Diastolic Blood Pressure Thresholds at Week 18
Description: number of participants achieving seated systolic and diastolic blood pressure thresholds BP<135/85, BP<130/80, BP<125/75, BP<120/80, SBP<135, SBP<130, SBP<125, SBP<120, DBP<85, DBP<80, DBP<75 at week 18
Time Frame: week 0 - week 18
Measure: Number; unit: participants
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 164
participants
  mean BP < 135/85 | 117
  mean BP < 130/80 | 87
  mean BP < 125/75 | 56
  mean BP < 120/80 | 49
  mean SBP < 135 | 123
  mean SBP < 130 | 101
  mean SBP < 125 | 74
  mean SBP < 120 | 51
  mean DBP < 85 | 147
  mean DBP < 80 | 128
  mean DBP < 75 | 94

18. Secondary Outcome: Number of Participants Achieving Mean 24 Hour Ambulatory Systolic and Diastolic Blood Pressure Reductions at Week 12
Description: number of participants achieving mean 24 hour ambulatory systolic and diastolic blood pressure reductions of; SBP reduction <= 15 mmHg, SBP reduction > 15 mmHg & <= 30 mmHg, SBP reduction > 30 mmHg & <= 45 mmHg, SBP reduction > 45 mmHg, DBP reduction <= 10 mmHg, DBP reduction > 10 mmHg & <= 15 mmHg, DBP reduction > 15 mmHg & <= 20 mmHg, DBP reduction > 20 mmHg at week 12
Time Frame: week 0 - week 12
Measure: Number; unit: participants
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 165
participants
  mean 24-hour SBP reduction =<15 mm Hg | 50
  mean 24-hour SBP reduction >15 & =<30 mm Hg | 91
  mean 24-hour SBP reduction >30 & =<45 mm Hg | 22
  mean 24-hour SBP reduction >45 mm Hg | 2
  mean 24-hour DBP reduction =<10 mm Hg | 72
  mean 24-hour DBP reduction >10 & =<15 mm Hg | 47
  mean 24-hour DBP reduction >15 & =<20 mm Hg | 31
  mean 24-hour DBP reduction >20 mm Hg | 15

19. Secondary Outcome: Number of Participants Achieving Mean Daytime Ambulatory Systolic and Diastolic Blood Pressure Reductions at Week 12
Description: number of participants achieving mean daytime ambulatory systolic and diastolic blood pressure reductions of; SBP reduction <= 15 mmHg, SBP reduction > 15 mmHg & <= 30 mmHg, SBP reduction > 30 mmHg & <= 45 mmHg, SBP reduction > 45 mmHg, DBP reduction <= 10 mmHg, DBP reduction > 10 mmHg & <= 15 mmHg, DBP reduction > 15 mmHg & <= 20 mmHg, DBP reduction > 20 mmHg at week 12
Time Frame: week 0 - week 12
Measure: Number; unit: participants
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 165
participants
  mean daytime SBP reduction =<15 mm Hg | 47
  mean daytime SBP reduction >15 & =<30 mm Hg | 84
  mean daytime SBP reduction >30 & =<45 mm Hg | 31
  mean daytime SBP reduction >45 mm Hg | 3
  mean daytime DBP reduction =<10 mm Hg | 68
  mean daytime DBP reduction >10 & =<15 mm Hg | 41
  mean daytime DBP reduction >15 & =<20 mm Hg | 33
  mean daytime DBP reduction >20 mm Hg | 23

20. Secondary Outcome: Number of Participants Achieving Mean Nighttime Ambulatory Systolic and Diastolic Blood Pressure Reductions at Week 12
Description: number of participants achieving mean nighttime ambulatory systolic and diastolic blood pressure reductions of; SBP reduction <= 15 mmHg, SBP reduction > 15 mmHg & <= 30 mmHg, SBP reduction > 30 mmHg & <= 45 mmHg, SBP reduction > 45 mmHg, DBP reduction <= 10 mmHg, DBP reduction > 10 mmHg & <= 15 mmHg, DBP reduction > 15 mmHg & <= 20 mmHg, DBP reduction > 20 mmHg at week 12
Time Frame: week 0 - week 12
Measure: Number; unit: participants
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 165
participants
  mean nighttime SBP reduction =<15 mm Hg | 60
  mean nighttime SBP reduction >15 & =<30 mm Hg | 79
  mean nighttime SBP reduction >30 & =<45 mm Hg | 21
  mean nighttime SBP reduction >45 mm Hg | 5
  mean nighttime DBP reduction =<10 mm Hg | 80
  mean nighttime SBP reduction >10 & =<15 mm Hg | 41
  mean nighttime SBP reduction >15 & =<20 mm Hg | 21
  mean nighttime DBP reduction >20 mm Hg | 23

21. Secondary Outcome: Number of Participants Achieving Mean Last 6 Hour Ambulatory Systolic and Diastolic Blood Pressure Reductions at Week 12
Description: number of participants achieving mean last 6 hour ambulatory systolic and diastolic blood pressure reductions of; SBP reduction <= 15 mmHg, SBP reduction > 15 mmHg & <= 30 mmHg, SBP reduction > 30 mmHg & <= 45 mmHg, SBP reduction > 45 mmHg, DBP reduction <= 10 mmHg, DBP reduction > 10 mmHg & <= 15 mmHg, DBP reduction > 15 mmHg & <= 20 mmHg, DBP reduction > 20 mmHg at week 12
Time Frame: week 0 - week 12
Measure: Number; unit: participants
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 165
participants
  mean last 6 hour SBP reduction =<15 mm Hg | 61
  mean last 6 hour SBP reduction >15 & =<30 mm Hg | 76
  mean last 6 hour SBP reduction >30 & =<45 mm Hg | 23
  mean last 6 hour SBP reduction >45 mm Hg | 5
  mean last 6 hour DBP reduction =<10 mm Hg | 76
  mean last 6 hour DBP reduction >10 & =<15 mm Hg | 41
  mean last 6 hour DBP reduction >15 & =<20 mm Hg | 27
  mean last 6 hour DBP reduction >20 mm Hg | 21

22. Secondary Outcome: Number of Participants Achieving Mean Last 4 Hour Ambulatory Systolic and Diastolic Blood Pressure Reductions
Description: number of participants achieving mean last 4 hour ambulatory systolic and diastolic blood pressure reductions of; SBP reduction <= 15 mmHg, SBP reduction > 15 mmHg & <= 30 mmHg, SBP reduction > 30 mmHg & <= 45 mmHg, SBP reduction > 45 mmHg, DBP reduction <= 10 mmHg, DBP reduction > 10 mmHg & <= 15 mmHg, DBP reduction > 15 mmHg & <= 20 mmHg, DBP reduction > 20 mmHg at week 12
Time Frame: week 0 - week 12
Measure: Number; unit: participants
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 165
participants
  mean last 4 hour SBP reduction =<15 mm Hg | 67
  mean last 4 hour SBP reduction >15 & =<30 mm Hg | 65
  mean last 4 hour SBP reduction >30 & =<45 mm Hg | 28
  mean last 4 hour SBP reduction >45 mm Hg | 5
  mean last 4 hour DBP reduction =<10 mm Hg | 76
  mean last 4 hour DBP reduction >10 & =<15 mm Hg | 36
  mean last 4 hour DBP reduction >15 & =<20 mm Hg | 25
  mean last 4 hour DBP reduction >20 mm Hg | 28

23. Secondary Outcome: Number of Participants Achieving Mean Last 2 Hour Ambulatory Systolic and Diastolic Blood Pressure Reductions at Week 12
Description: number of participants achieving mean last 2 hour ambulatory systolic and diastolic blood pressure reductions of; SBP reduction <= 15 mmHg, SBP reduction > 15 mmHg & <= 30 mmHg, SBP reduction > 30 mmHg & <= 45 mmHg, SBP reduction > 45 mmHg, DBP reduction <= 10 mmHg, DBP reduction > 10 mmHg & <= 15 mmHg, DBP reduction > 15 mmHg & <= 20 mmHg, DBP reduction > 20 mmHg at week 12
Time Frame: week 0 - week 12
Measure: Number; unit: participants
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 165
participants
  mean last 2 hour SBP reduction =<15 mm Hg | 63
  mean last 2 hour SBP reduction >15 & =<30 mm Hg | 62
  mean last 2 hour SBP reduction >30 & =<45 mm Hg | 35
  mean last 2 hour SBP reduction >45 mm Hg | 5
  mean last 2 hour DBP reduction =<10 mm Hg | 77
  mean last 2 hour DBP reduction >10 & =<15 mm Hg | 28
  mean last 2 hour DBP reduction >15 & =<20 mm Hg | 29
  mean last 2 hour DBP reduction >20 mm Hg | 31

24. Secondary Outcome: Number of Participants Achieving Mean Seated Systolic and Diastolic Blood Pressure Reductions at Week 3
Description: number of participants achieving mean seated systolic and diastolic blood pressure reductions of; SBP reduction <= 15 mmHg, SBP reduction > 15 mmHg & <= 30 mmHg, SBP reduction > 30 mmHg & <= 45 mmHg, SBP reduction > 45 mmHg, DBP reduction <= 10 mmHg, DBP reduction > 10 mmHg & <= 15 mmHg, DBP reduction > 15 mmHg & <= 20 mmHg, DBP reduction > 20 mmHg at week 3
Time Frame: week 0 - week 3
Measure: Number; unit: participants
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 201
participants
  mean seated SBP reduction =<15 mm Hg | 131
  mean seated SBP reduction >15 & =<30 mm Hg | 62
  mean seated SBP reduction >30 & =<45 mm Hg | 6
  mean seated SBP reduction >45 mm Hg | 2
  mean seated DBP reduction =<10 mm Hg | 163
  mean seated DBP reduction >10 & =<15 mm Hg | 25
  mean seated DBP reduction >15 & =<20 mm Hg | 10
  mean seated DBP reduction >20 mm Hg | 3

25. Secondary Outcome: Number of Participants Achieving Mean Seated Systolic and Diastolic Blood Pressure Reductions at Week 6
Description: number of participants achieving mean seated systolic and diastolic blood pressure reductions of; SBP reduction <= 15 mmHg, SBP reduction > 15 mmHg & <= 30 mmHg, SBP reduction > 30 mmHg & <= 45 mmHg, SBP reduction > 45 mmHg, DBP reduction <= 10 mmHg, DBP reduction > 10 mmHg & <= 15 mmHg, DBP reduction > 15 mmHg & <= 20 mmHg, DBP reduction > 20 mmHg at week 6
Time Frame: week 0 - week 6
Measure: Number; unit: participants
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 192
participants
  mean seated SBP reduction =<15 mm Hg | 69
  mean seated SBP reduction >15 & =<30 mm Hg | 90
  mean seated SBP reduction >30 & =<45 mm Hg | 31
  mean seated SBP reduction >45 mm Hg | 2
  mean seated DBP reduction =<10 mm Hg | 120
  mean seated DBP reduction >10 & =<15 mm Hg | 33
  mean seated DBP reduction >15 & =<20 mm Hg | 24
  mean seated DBP reduction >20 mm Hg | 15

26. Secondary Outcome: Number of Participants Achieving Mean Seated Systolic and Diastolic Blood Pressure Reductions at Week 9
Description: number of participants achieving mean seated systolic and diastolic blood pressure reductions of; SBP reduction <= 15 mmHg, SBP reduction > 15 mmHg & <= 30 mmHg, SBP reduction > 30 mmHg & <= 45 mmHg, SBP reduction > 45 mmHg, DBP reduction <= 10 mmHg, DBP reduction > 10 mmHg & <= 15 mmHg, DBP reduction > 15 mmHg & <= 20 mmHg, DBP reduction > 20 mmHg at week 9
Time Frame: week 0 - week 9
Measure: Number; unit: participants
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 184
participants
  mean seated SBP reduction =<15 mm Hg | 72
  mean seated SBP reduction >15 & =<30 mm Hg | 69
  mean seated SBP reduction >30 & =<45 mm Hg | 34
  mean seated SBP reduction >45 mm Hg | 9
  mean seated DBP reduction =<10 mm Hg | 100
  mean seated DBP reduction >10 & =<15 mm Hg | 43
  mean seated DBP reduction >15 & =<20 mm Hg | 18
  mean seated DBP reduction >20 mm Hg | 23

27. Secondary Outcome: Number of Participants Achieving Mean Seated Systolic and Diastolic Blood Pressure Reductions at Week 12
Description: number of participants achieving mean seated systolic and diastolic blood pressure reductions of; SBP reduction <= 15 mmHg, SBP reduction > 15 mmHg & <= 30 mmHg, SBP reduction > 30 mmHg & <= 45 mmHg, SBP reduction > 45 mmHg, DBP reduction <= 10 mmHg, DBP reduction > 10 mmHg & <= 15 mmHg, DBP reduction > 15 mmHg & <= 20 mmHg, DBP reduction > 20 mmHg at week 12
Time Frame: week 0 - week 12
Measure: Number; unit: participants
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 177
participants
  mean seated SBP reduction =<15 mm Hg | 48
  mean seated SBP reduction >15 & =<30 mm Hg | 73
  mean seated SBP reduction >30 & =<45 mm Hg | 45
  mean seated SBP reduction >45 mm Hg | 11
  mean seated DBP reduction =<10 mm Hg | 85
  mean seated DBP reduction >10 & =<15 mm Hg | 42
  mean seated DBP reduction >15 & =<20 mm Hg | 27
  mean seated DBP reduction >20 mm Hg | 23

28. Secondary Outcome: Number of Participants Achieving Mean Seated Systolic and Diastolic Blood Pressure Reductions at Week 15
Description: number of participants achieving mean seated systolic and diastolic blood pressure reductions of; SBP reduction <= 15 mmHg, SBP reduction > 15 mmHg & <= 30 mmHg, SBP reduction > 30 mmHg & <= 45 mmHg, SBP reduction > 45 mmHg, DBP reduction <= 10 mmHg, DBP reduction > 10 mmHg & <= 15 mmHg, DBP reduction > 15 mmHg & <= 20 mmHg, DBP reduction > 20 mmHg at week 15
Time Frame: week 0 - week 15
Measure: Number; unit: participants
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 172
participants
  mean seated SBP reduction =<15 mm Hg | 31
  mean seated SBP reduction >15 & =<30 mm Hg | 66
  mean seated SBP reduction >30 & =<45 mm Hg | 55
  mean seated SBP reduction >45 mm Hg | 20
  mean seated DBP reduction =<10 mm Hg | 52
  mean seated DBP reduction >10 & =<15 mm Hg | 45
  mean seated DBP reduction >15 & =<20 mm Hg | 32
  mean seated DBP reduction >20 mm Hg | 43

29. Secondary Outcome: Number of Participants Achieving Mean Seated Systolic and Diastolic Blood Pressure Reductions at Week 18
Description: number of participants achieving mean seated systolic and diastolic blood pressure reductions of; SBP reduction <= 15 mmHg, SBP reduction > 15 mmHg & <= 30 mmHg, SBP reduction > 30 mmHg & <= 45 mmHg, SBP reduction > 45 mmHg, DBP reduction <= 10 mmHg, DBP reduction > 10 mmHg & <= 15 mmHg, DBP reduction > 15 mmHg & <= 20 mmHg, DBP reduction > 20 mmHg at week 18
Time Frame: week 0 - week 18
Measure: Number; unit: participants
Arm/Group | Aml + Olm + Hctz
Number analyzed (Participants) | 164
participants
  mean seated SBP reduction =<15 mm Hg | 22
  mean seated SBP reduction >15 & =<30 mm Hg | 53
  mean seated SBP reduction >30 & =<45 mm Hg | 64
  mean seated SBP reduction >45 mm Hg | 25
  mean seated DBP reduction =<10 mm Hg | 50
  mean seated DBP reduction >10 & =<15 mm Hg | 33
  mean seated DBP reduction >15 & =<20 mm Hg | 29
  mean seated DBP reduction >20 mm Hg | 52

ADVERSE EVENTS:
Groups:
- ALL - Aml + Olm + Hctz: Summary of ALL participants receiving amlodipine + olmesartan medoxomil, if required, + hydrochlorothiazide, if required
- Start - Amlodipine 5 mg: All participants started trial on Amlodipine 5 mg.
- Titration 1 - Amlodipine 5 mg / Olmesartan 20 mg; Titration 2 - Amlodipine 5 mg / Olmesartan 40 mg; Titration 3 - Amlodipine 10 mg / Olmesartan 40 mg; Titration 4 Amlodipine 10 mg / Olmesartan 40 mg / HCTZ 12.5 mg; Titration 5 - Amlodipine 10 mg / Olmesartan 40 mg / HCTZ 25 mg: Participants not meeting blood pressure (BP) goals on previous regimen were titrated to this regimen.
Arm/Group | ALL - Aml + Olm + Hctz | Start - Amlodipine 5 mg | Titration 1 - Amlodipine 5 mg / Olmesartan 20 mg | Titration 2 - Amlodipine 5 mg / Olmesartan 40 mg | Titration 3 - Amlodipine 10 mg / Olmesartan 40 mg | Titration 4 Amlodipine 10 mg / Olmesartan 40 mg / HCTZ 12.5 mg | Titration 5 - Amlodipine 10 mg / Olmesartan 40 mg / HCTZ 25 mg
Serious Adverse Events (participants affected / at risk) | 4/207 | 0/207 | 0/195 | 1/177 | 0/167 | 1/146 | 2/101
Other Adverse Events (participants affected / at risk) | 80/207 | 16/207 | 15/195 | 10/177 | 21/167 | 14/146 | 4/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALL - Aml + Olm + Hctz (N=207) | Start - Amlodipine 5 mg (N=207) | Titration 1 - Amlodipine 5 mg / Olmesartan 20 mg (N=195) | Titration 2 - Amlodipine 5 mg / Olmesartan 40 mg (N=177) | Titration 3 - Amlodipine 10 mg / Olmesartan 40 mg (N=167) | Titration 4 Amlodipine 10 mg / Olmesartan 40 mg / HCTZ 12.5 mg (N=146) | Titration 5 - Amlodipine 10 mg / Olmesartan 40 mg / HCTZ 25 mg (N=101)
pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALL - Aml + Olm + Hctz (N=207) | Start - Amlodipine 5 mg (N=207) | Titration 1 - Amlodipine 5 mg / Olmesartan 20 mg (N=195) | Titration 2 - Amlodipine 5 mg / Olmesartan 40 mg (N=177) | Titration 3 - Amlodipine 10 mg / Olmesartan 40 mg (N=167) | Titration 4 Amlodipine 10 mg / Olmesartan 40 mg / HCTZ 12.5 mg (N=146) | Titration 5 - Amlodipine 10 mg / Olmesartan 40 mg / HCTZ 25 mg (N=101)
anaemia (Blood and lymphatic system disorders) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 2 (2)
oedema peripheral (General disorders) | 20 (20) | 7 (7) | 3 (3) | 2 (2) | 7 (7) | 1 (1) | 0 (0)
upper respiratory tract infection (Infections and infestations) | 11 (11) | 0 (0) | 2 (2) | 3 (3) | 3 (3) | 3 (3) | 0 (0)
bronchitis (Infections and infestations) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
dizziness (Nervous system disorders) | 12 (12) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 5 (5) | 0 (0)
headache (Nervous system disorders) | 6 (6) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
hypotension (Vascular disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reflects the following restrictive language in the Clinical Study Agreements: "If identified by Daiichi Sankyo Inc. (DSI), any of DSI's confidential information as defined herein shall be deleted. Nothing in this publication section shall be taken as giving DSI any right of editorial control over any publication prepared by the Study Site."